CLINICAL TRIAL: NCT05038410
Title: Randomized, Double-blind, Placebo-controlled, Crossover Study to Investigate the Mechanism of Action of an Oral Enzyme Treatment With Bromelain, Trypsin and Rutoside Versus Placebo in Subjects With OsTeoarthritis
Brief Title: Study to Investigate the Mechanism of Action of an Oral Enzyme Treatment With Bromelain, Trypsin and Rutoside Versus Placebo in Subjects With OsTeoarthritis
Acronym: WobeSmart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mucos Pharma GmbH & Co. KG (Industry)
Collaborators: Société des Produits Nestlé (SPN) (Industry); Artialis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020CLI
Record Dates: First submitted 2021-05-25; First posted 2021-09-09 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Wobenzym

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wobenzym® (Active Comparator): Medicinal product Wobenzym® containing Bromelain (67.5-76.5 mg) adjusted to 450 FIP units, Trypsin (32-48mg) adjusted to 24 µkat and Rutoside trihydrate (100mg).
  Interventions: Drug: Wobenzym®
- PLACEBO (Placebo Comparator): No active ingredients. The active ingredients will be substituted by microcrystalline cellulose.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Wobenzym® — Wobenzym®
  Arms: Wobenzym®
Other: Placebo — Microcrystalline cellulose
  Arms: PLACEBO

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamic profile of an oral enzyme treatment with Bromelain, Trypsin and Rutoside in subjects with osteoarthritis.

DETAILED DESCRIPTION:
This study is a randomised, placebo controlled, two parallel arms, cross over, and multicentric trial in 40 male and female subjects suffering from osteoarthritis. While is it well established that Wobenzyme is safe and have proven efficacy in painful conditions, inflammation and osteoarthritis, little is known about its clear mechanism of action underlying its clinical efficacy. This study hypothesises that oral enzyme combination therapy with Wobenzyme will lead to systemic pharmacodynamic effects which will be documented by a holistic assessment of the inflammasome, innate immune system, cartilage turnover, systemic inflammatory markers, as well as potential cellular pathways.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 40 years of age and with BMI ≤ 35 kg/m2;
2. Uni- or bilateral femorotibial knee OA :

   1. Responding to clinical and radiological criteria of American College of Rheumatology (ACR);
   2. Symptomatic for more than 6 months in the index knee;
   3. Radiological Kellgren & Lawrence (K&L) grade II-III in standing x-rays from less than 12 months.
3. Mild-to-Moderate mean knee pain score at rest or at walking over the last 24 hours on the index knee evaluated on VAS (0-100) ≥ 40 at baseline;
4. Able to follow the instructions of the study;
5. Having signed an informed consent.

Exclusion Criteria:

Related to knee:

1. Recent macro-trauma of the knee responsible of the symptomatic knee left to the Investigator's discretion;
2. Concurrent articular disease interfering with the evaluation of pain left to the Investigator's discretion;
3. Prosthesis in the target knee;
4. Knee swelling requiring corticosteroids local injection.

   Related to treatments:
5. Analgesics to manage knee pain 24 hours before inclusion visit;
6. Corticosteroids injection in the target knee in the last 3 months;
7. Hyaluronan injection in the target knee in the last 6 months;
8. Arthroscopy in the last 6 months;
9. Oral corticotherapy ≥ 5mg/day (in Prednisolone equivalent) in the last 3 months;
10. Symptomatic slow-acting drugs for osteoarthritis (SYSADOA) or dietary supplement, i.e., curcuma extract, chondroitin, glucosamine, diacerein or avocado-soya unsaponifiables in the last 3 months;
11. An anticipated need for any forbidden treatments during the trial;
12. Contraindications to the product :

    1. severe hepatic and renal impairment
    2. congenital or acquired coagulation disorders, e.g. haemophilia
    3. severe liver and/or kidney damage
    4. hereditary galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
13. Hypersensitivity or allergy to the product components, and pineapple;
14. Treatments based on strontium ranelate, bisphosphonates, selective estrogen-receptor modulator (SERM) and parathormone (PTH) in the last 12 months;
15. Treatment based on zoledronate in the last 2 years;
16. Treatment based on denosumab in the last 6 months;
17. Treatment with anticoagulants and/or anti-platelet agents

    Related to associated diseases:
18. Any severe, uncontrolled and limiting disease left to the Investigator's discretion;
19. Patient with widespread pain/depression (e.g. fibromyalgia);
20. Lower or upper extremity surgery or fracture in the last 6 months;
21. Anticipated need for any surgical or other invasive procedure during the trial including prosthesis in the target knee;
22. Severe alteration of mobility enabling functional evaluation.

    Related to subjects
23. Close collaborators to the investigational team, the study coordinator (ARTIALIS) or to the Sponsor;
24. Currently participating or having participated in another therapeutic clinical trial in the three previous months;
25. Having made a blood donation in the past month;
26. Under guardianship or judicial protection;
27. Pregnancy, breastfeeding, planned conception, or premenopausal women without effective contraception (tablet, patch, ring, diaphragm, implant and intrauterine device, tubal ligation or hysterectomy);
28. Counter-indication to an MRI examination.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Effects on cartilage biomarkers | 20 weeks
  Change in sera biomarkers sColl2-1, sColl2-1NO2, sCOMP, sPIIANP and urine biomarker uCTXII between visit 0 and visit 5 measured using immunoassays (Enzyme-linked Immunosorbent assay, ELISA)
Effects on markers of innate immune response | 20 weeks
  Change in the expression of M1/M2 Polarization specific membrane markers on fresh blood macrophage, between visit 0 and visit 5 using flow cytometry
Effects on systemic inflammatory markers | 20 weeks
  Change in sera biomarkers NLRP 3 Inflammasome, α-2-macroglobulin, IL-1β, TNFα, IL-6, IL-10, IL-4 between visit 0 and visit 5 measured using immunoassays (Enzyme-linked Immunosorbent assay, ELISA)
Effects on cellular pathways | 20 weeks
  Change in plasma proteomic profile using liquid chromatography-tandem mass spectrometry (LC-MS/MS) between visit 0 and visit 5.

SECONDARY OUTCOMES:
Vital signs and anthropomorphic measurements | 40 weeks
  Changes in systolic and diastolic Blood pressure (BP) in mmHg between visit -1 and visit 6
Vital signs and anthropomorphic measurements | 40 weeks
  Changes in Heart Rate (HR) measured in beats per minute between visit -1 and visit 6
Vital signs and anthropomorphic measurements | 40 weeks
  Changes in Temperature measured in degrees Celsius between visit -1 and visit 6
Vital signs and anthropomorphic measurements | 40 weeks
  Changes in weight measured in kilograms, height measured in centimeters and BMI (weight and height will be combined to calculate BMI in kg/m2 between visit -1 and visit 6
Knee Pain | 36 weeks
  Changes in knee pain at rest and while walking using a Visual Analogue Scale (1 to 100 mm scale where a higher score indicates greater pain intensity) between visit 0 and visit 6
Knee Function | 36 weeks
  Changes in knee function using Knee injury and Osteoarthristis Outcome Score (KOOS). KOOS is a self-administrated questionnaire comprising 5 subscales: pains, symptoms, activities of daily living, sports and recreation function, and quality of life (0 to 100 scale where 100 indicates the best result) between visit 0 and visit 6
Patient global assessment of disease activity (PGADA) | 36 weeks
  Changes in PGADA using a Visual Analogue Scale (1 to 100 mm scale where a higher score indicates a higher level of disease activity /a worse global health) between visit 0 and visit 6
Patient physical activity | 36 weeks
  Effects on subject mobility using a connected device to record heart rate (beats/min between visit 0 and visit 6
Patient physical activity | 36 weeks
  Effects on subject mobility using a connected device to record number of steps/day taken between visit 0 and visit 6
Patient physical activity | 36 weeks
  Effects on subject mobility using a connected device to record number of climbed stairs/day between visit 0 and visit 6
Patient physical activity | 36 weeks
  Effects on subject mobility using a connected device to record intensive exercise minutes/day between visit 0 and visit 6
Patient physical activity | 36 weeks
  Effects on subject mobility using a connected device to record calories burned/day between visit 0 and visit 6minutes/day between visit 0 and visit 6
Body metabolism | 20 weeks
  Effects on body metabolism marker TGF-β1, TGF β 2, TGF-β 3 using immunoassays (Enzyme-linked Immunosorbent assay, ELISA) between visit 0 and visit 5
Clinical chemistry | 20 weeks
  Number of participants with changes in clinical chemistry measurements (concentration of myostatin, hemoglobin, hematocrit, erythrocyte count, TG, TC, LDL, HDL, glucose, hsCRP, uric acid, coagulation markers and key hepatic enzymes) using immunoassays between visit 0 and visit 5
Joint structure modification | 36 weeks
  Effects on joint structure using either MRI Osteoarthritis Knee Score (MOAKS - a semi quantitative scoring tool. Fourteen subregions are defined for scoring of articular cartilage and bone marrow lesions from grade 0 to grade 3. The more the grade increases, the more important the pathology) or Whole-Organ Magnetic Resonance Imaging Score (WORMS - a semi quantitative scoring tool that examines a spectrum of OA-related structural abnormalities including soft tissue, cartilage and bone in the knee at various anatomical subregion locations. The more the score increases, the more important the pathology) between visit 0 and visit 6
Volume of joint effusion | 36 weeks
  Volume of joint effusion by MRI using volumetric segmentation method between visit 0 and visit 6
Tolerance | 40 weeks
  Number of patients with Adverse Events, type of reported adverse events and subject drop out between visit -1 and visit 6
Compliance | 36 weeks
  Tablet count of investigational product between visit 0 and visit 6
Responder rate to treatment | 36 weeks
  Responder rate to treatment defined as changes in knee pain and/or knee function and/or patients disease activity using Pain and/or PGADA and/or KOOS according to recommendations of OMERACT OARSI (Osteoarthritis Research Society International (OARSI) Standing Committee for Clinical Trials Response Criteria Initiative and the Outcome Measures in Rheumatology (OMERACT), defined by either a high improvement in pain or in function >50% and absolute change >20 or an improvement in at least 2 of the 3 following: pain >20% and absolute change >10, function >20% and absolute change >10, patient's global assessment >20% and absolute change >10 (between visit 0 and visit 6

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Badot, Principal Investigator — Centre Hospitalier Universitaire (CHU) Brugmann; Didier Urbin-Choffray, Principal Investigator — Centre Hospitalier Regional de la Citadelle; Karl Brabants, Principal Investigator — Ziekenhuis Netwerk Antwerpen (ZNA) Middelheim; Jean-Emile Dubuc, Principal Investigator — Cliniques Universitaires Saint Luc UCL; Siddhartha Lieten, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (5):
- Belgium (5):
  - Ziekenhuis Netwerk Antwerpen (ZNA) Middelheim, Antwerp
  - Centre Hospitalier Universitaire (CHU) Brugmann, Brussels
  - Cliniques Universitaires Saint Luc UCL, Brussels
  - UZ Brussel, Jette
  - Centre Hospitalier Régional de la Citadelle, Liège

REFERENCES:
- [Derived] Henrotin Y, Pap T, Lieten S, Badot V, Dubuc JE, Urbin-Choffray D, von Eynatten M, Johansen OE, Rau S, Brabants K. Oral enzyme combination therapy reduces systemic inflammation, urinary CTXII and pain in knee osteoarthritis: a proof-of-mechanism, randomised, crossover, double-blind, placebo-controlled trial. RMD Open. 2025 Aug 12;11(3):e005433. doi: 10.1136/rmdopen-2025-005433. PMID 40803821